CLINICAL TRIAL: NCT05353933
Title: Efficacy and Safety of Thread Embedding Acupuncture Combined With PPI in Treating GERD
Brief Title: Efficacy and Safety of Thread Embedding Acupuncture in Treating Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 606/HDDD-DHYD
Record Dates: First submitted 2022-04-16; First posted 2022-04-29 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator who examine GERD-related symptoms and outcome assessor will be blinded.
  However, the investigator who examine the side effects of thread embedding acupuncture will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEA + PPI (Experimental): Thread embedding acupuncture (TEA) every 2 weeks in 4 weeks (twice). Combined with oral pantoprazole 40 mg capsules (Pantostad 40 CAP) once daily for 4 weeks.
  Interventions: Other: Thread embedding acupuncture; Drug: Pantoprazole 40mg
- PPI (Active Comparator): Oral pantoprazole 40 mg capsules (Pantostad 40 CAP) once daily for 4 weeks.
  Interventions: Drug: Pantoprazole 40mg

INTERVENTIONS:
Other: Thread embedding acupuncture — Thread embedding acupuncture (TEA) that use chromic catgut thread with 3/0 size with 1 centimeter long for each acupoint (TRUSTIGUT® (C), CPT Sutures Co., Ltd, Ho Chi Minh, Vietnam). Every 2 weeks in 4 weeks (twice), 13 acupoints will be embedded including Xiawan (CV-10), Zhongwan (CV-12), Shangwan (CV-13) and Zusanli (ST-36), Neiguan (PC-6), Geshu (BL-17), Ganshu (BL-18), Pishu (BL-20) in both sides of the body.
  Arms: TEA + PPI
Drug: Pantoprazole 40mg — Oral pantoprazole 40 mg capsules (Pantostad 40 CAP, Stellapharm J.V. Co., Ltd, Binh Duong, Vietnam) thirty minutes to one hour before the first meal once daily for 4 weeks.

SUMMARY:
Gastroesophageal reflux disease is a very common disease nowadays. Proton-pump inhibitors (PPIs) are the first-line treatment for this disease. However, the effectiveness of treatment with PPIs is still limited. Acupuncture has been shown to be effective in treating this condition. Another treatment method is thread embedding acupuncture therapy, which is a method of burying threads into acupoints to create a more lasting stimulation than traditional acupuncture.

This study will evaluate the efficacy and safety of the combination of thread embedding acupuncture and standard dose pantoprazole compared with standard dose pantoprazole as monotherapy in adults.

DETAILED DESCRIPTION:
Patients with GERD diagnosed based on the GerdQ score who meet the inclusion criteria and do not meet the exclusion criteria will be included in the study. After randomization, patients will be divided into 2 groups: control group and intervention group. In both groups, patients will be treated for GERD according to current guidelines including PPIs, additional antacids as needed, and lifestyle changes. The intervention group will include additional thread embedding acupuncture therapy (TEA) twice on day 0 and day 14th. Intervention duration is 4 weeks.

The objectives of the study are to evaluate the improvement of GERD symptoms by using the evaluation score including Gastroesophageal reflux disease questionnaire (GerdQ) and Frequency Scale for the Symptoms of GERD (FSSG); the evaluation score of Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) will be used to evaluate the improvement of quality of life; and evaluate the safety of TEA in the treatment of GERD.

All scales will be evaluated before and after the intervention. For the GerdQ score, patients will be assessed weekly, every 2 weeks for FSSG and GERD-HRQL during the 4-week intervention. For TEA's side effects, it will be assessed regularly during the 4-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-60 years of age.
* Patients with total scores ≥ 8 on the Gastroesophageal Reflux Disease Questionnaire (GerdQ) and scores ≥ 2 for each symptom including heartburn and/or regurgitation.
* Ability to read, understand and provide informed consent.
* Currently not receiving any intervention to treat GERD.

Exclusion Criteria:

* Have any current symptoms related to a structural disease that has been confirmed by endoscopy (e.g., gastrointestinal cancer, eosinophilic esophagitis, candida esophagitis, peptic ulcers, Zollinger-Ellison syndrome, pyloric stenosis, etc.).
* With known inflammatory bowel disease or other serious disease (hepatic, renal, respiratory, or cardiac disease) or rare genetic diseases (such as fructose intolerance, glucose-galactose malabsorption, saccharose-isomaltose deficiency), severe concomitant diseases, or a history of alcohol or drug abuse.
* Have severe dysphagia, hematemesis, weight loss, or hematochezia.
* A history of oesophageal and/or gastrointestinal surgery.
* Current use of drugs affecting treatment and evaluation of GERD including systemic glucocorticoids, nonsteroidal anti-inflammatory, calcium channel blockers, anticholinergics, bisphosphonates, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, tetracycline, HIV protease inhibitors, rifampin, potassium supplements, iron, quinidine, zidovudine, anticholinergic agents, alpha-adrenergic antagonists, β2-adrenergic agonists, benzodiazepines, barbiturates, dopamine, estrogens, progesterone, narcotic analgesics, nitrates, prostaglandins, theophylline.
* Are being treated with proton-pump inhibitors within the last 14 days, H2-receptor antagonists, or prokinetics within the last 10 days, intake of alginates or antacids within the last 3 days or using any traditional medicine to treat GERD within the last 2 weeks.
* A history of hypersensitivity reaction with PPIs (including their components), catgut or acupuncture or thread embedding acupuncture treatment.
* Are pregnant or breastfeeding.
* Are taking part in any other clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in the Gastroesophageal reflux disease questionnaire score (GerdQ) after each week of treatment. | Assessments at day 0 and after every week during 4-week treatment (day 7th, day 14th, day 21st, day 28th).
  According to GerdQ, patients were asked to reflect on their symptoms and use of over-the-counter medications over the preceding week. It uses a four graded Likert scale (0-3) to score giving a total GerdQ score range of 0-18. High score indicates serious disease.
Change in the proportion of GERD typical symptoms absence after each week of treatment. | Assessments at day 0 and after every week during 4-week treatment (day 7th, day 14th, day 21st, day 28th).
  Based on the GerdQ score, when the answers for questions 1 and 2 are zero, the disappearance of typical symptoms including heartburn and regurgitation respectively will be determined.

SECONDARY OUTCOMES:
Change in the GERD symptoms frequency after every two weeks of treatment. | Assessments day 0 and every two weeks during 4-week treatment (day 14th, day 28th).
  GERD symptoms frequency will be assessed by the Frequency Scale for the Symptoms of GERD (FSSG). The FSSG questionnaire comprises twelve questions in two domains, the reflux symptom domain and dysmotility symptom domain. The FSSG uses a 5-point Likert scale (0-4). Total FSSG score range of 0-48. High score indicates serious disease.
Change in the health related quality of life after every two weeks of treatment. | Assessments at day 0 and every two weeks during 4-week treatment (day 14th, day 28th).
  Health related quality of life will be assessed by the Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) instrument. The GERD-HRQL with 16 questions uses a numerical Likert-type response, whereby each patient assesses the severity of symptoms on an ordinal scale (0-5). The GERD-HRQL has a possible range of 0-80, with the heartburn, regurgitation and other arms. High score indicates serious disease.
The proportion of thread embedding acupuncture side effects. | Up to 4 weeks.
  TEA side effects include: post-treatment discomfort, post-treatment body temperature rising, local hematoma or subcutaneous hemorrhage, local swelling, local induration, local pain, local redness, infection, abscess, pruritus, anaphylaxis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Sakurai K, Suda H, Fujie S, Takeichi T, Okuda A, Murao T, Hasuda K, Hirano M, Ito K, Tsuruta K, Hattori M. Short-Term Symptomatic Relief in Gastroesophageal Reflux Disease: A Comparative Study of Esomeprazole and Vonoprazan. Dig Dis Sci. 2019 Mar;64(3):815-822. doi: 10.1007/s10620-018-5365-0. Epub 2018 Nov 10. PMID 30415407
- [Background] Han G, Leem J, Lee H, Lee J. Electroacupuncture to treat gastroesophageal reflux disease: study protocol for a randomized controlled trial. Trials. 2016 May 17;17(1):246. doi: 10.1186/s13063-016-1371-8. PMID 27188910
- [Background] Scholten T, Gatz G, Hole U. Once-daily pantoprazole 40 mg and esomeprazole 40 mg have equivalent overall efficacy in relieving GERD-related symptoms. Aliment Pharmacol Ther. 2003 Sep 15;18(6):587-94. doi: 10.1046/j.1365-2036.2003.01745.x. PMID 12969085
- [Background] Wong BC, Kinoshita Y. Systematic review on epidemiology of gastroesophageal reflux disease in Asia. Clin Gastroenterol Hepatol. 2006 Apr;4(4):398-407. doi: 10.1016/j.cgh.2005.10.011. PMID 16616342
- [Background] El-Serag H, Becher A, Jones R. Systematic review: persistent reflux symptoms on proton pump inhibitor therapy in primary care and community studies. Aliment Pharmacol Ther. 2010 Sep;32(6):720-37. doi: 10.1111/j.1365-2036.2010.04406.x. PMID 20662774
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Fock KM, Talley N, Goh KL, Sugano K, Katelaris P, Holtmann G, Pandolfino JE, Sharma P, Ang TL, Hongo M, Wu J, Chen M, Choi MG, Law NM, Sheu BS, Zhang J, Ho KY, Sollano J, Rani AA, Kositchaiwat C, Bhatia S. Asia-Pacific consensus on the management of gastro-oesophageal reflux disease: an update focusing on refractory reflux disease and Barrett's oesophagus. Gut. 2016 Sep;65(9):1402-15. doi: 10.1136/gutjnl-2016-311715. Epub 2016 Jun 3. PMID 27261337
- [Background] Zhou Y, Ma HQ, Yang ZJ, Shao HT, Yue GL, Du GZ. [Comparative study on effect of electroacupuncture at lower he-sea point of stomach and he-sea matching front-mu points for gastroparesis]. Zhongguo Zhen Jiu. 2020 Sep 12;40(9):925-7. doi: 10.13703/j.0255-2930.20191025-k0002. Chinese. PMID 32959584
- [Background] Gyawali CP, Fass R. Management of Gastroesophageal Reflux Disease. Gastroenterology. 2018 Jan;154(2):302-318. doi: 10.1053/j.gastro.2017.07.049. Epub 2017 Aug 5. PMID 28827081
- [Background] Gyawali CP, Kahrilas PJ, Savarino E, Zerbib F, Mion F, Smout AJPM, Vaezi M, Sifrim D, Fox MR, Vela MF, Tutuian R, Tack J, Bredenoord AJ, Pandolfino J, Roman S. Modern diagnosis of GERD: the Lyon Consensus. Gut. 2018 Jul;67(7):1351-1362. doi: 10.1136/gutjnl-2017-314722. Epub 2018 Feb 3. PMID 29437910
- [Background] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151
- [Background] Gao L, Chen B, Zhang Q, Zhao T, Li B, Sha T, Zou J, Guo Y, Pan X, Guo Y. Acupuncture with different acupoint combinations for chemotherapy-induced nausea and vomiting: study protocol for a randomized controlled trial. BMC Complement Altern Med. 2016 Nov 8;16(1):441. doi: 10.1186/s12906-016-1425-1. PMID 27821107
- [Background] Shen J, Wenger N, Glaspy J, Hays RD, Albert PS, Choi C, Shekelle PG. Electroacupuncture for control of myeloablative chemotherapy-induced emesis: A randomized controlled trial. JAMA. 2000 Dec 6;284(21):2755-61. doi: 10.1001/jama.284.21.2755. PMID 11105182
- [Background] Ho CE, Goh YL, Zhao XX, Yu CY, Zhang C. GERD: An Alternative Perspective. Psychosomatics. 2016 Mar-Apr;57(2):142-51. doi: 10.1016/j.psym.2015.10.007. Epub 2015 Oct 26. PMID 26895729
- [Background] Hunt R, Armstrong D, Katelaris P, Afihene M, Bane A, Bhatia S, Chen MH, Choi MG, Melo AC, Fock KM, Ford A, Hongo M, Khan A, Lazebnik L, Lindberg G, Lizarzabal M, Myint T, Moraes-Filho JP, Salis G, Lin JT, Vaidya R, Abdo A, LeMair A; Review Team:. World Gastroenterology Organisation Global Guidelines: GERD Global Perspective on Gastroesophageal Reflux Disease. J Clin Gastroenterol. 2017 Jul;51(6):467-478. doi: 10.1097/MCG.0000000000000854. No abstract available. PMID 28591069
- [Background] Huo J, Zhao J, Yuan Y, Wang J. [Research status of the effect mechanism on catgut-point embedding therapy]. Zhongguo Zhen Jiu. 2017 Nov 12;37(11):1251-4. doi: 10.13703/j.0255-2930.2017.11.031. Chinese. PMID 29354967
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Quach DT, Pham QTT, Tran TLT, Vu NTH, Le QD, Nguyen DTN, Dang NLB, Le HM, Le NQ. Clinical characteristics and risk factors of gastroesophageal reflux disease in Vietnamese patients with upper gastrointestinal symptoms undergoing esophagogastroduodenoscopy. JGH Open. 2021 Mar 26;5(5):580-584. doi: 10.1002/jgh3.12536. eCollection 2021 May. PMID 34013058
- [Background] Shuai X, Xie P, Liu J, Xiang Y, Li J, Lan Y. Different effects of electroacupuncture on esophageal motility and serum hormones in cats with esophagitis. Dis Esophagus. 2008;21(2):170-5. doi: 10.1111/j.1442-2050.2007.00757.x. PMID 18269654
- [Background] Sun QH, Li TT, Huang MT, Wang MY, Xiao X, Bai XH. [Acupoint selection rules in treating gastroesophageal reflux disease with acupuncture in China based on data mining]. Zhongguo Zhen Jiu. 2020 Dec 12;40(12):1374-8. doi: 10.13703/j.0255-2930.20191107-0003. Chinese. PMID 33415885
- [Background] Wang C, Zhou DF, Shuai XW, Liu JX, Xie PY. Effects and mechanisms of electroacupuncture at PC6 on frequency of transient lower esophageal sphincter relaxation in cats. World J Gastroenterol. 2007 Sep 28;13(36):4873-80. doi: 10.3748/wjg.v13.i36.4873. PMID 17828819
- [Background] Wang XL, Lin GH, Xu N, Zeng JC, Xu DH, Wang SX. [Analysis of adverse reactions of acupoint catgut embedding therapy]. Zhongguo Zhen Jiu. 2020 Feb 12;40(2):193-6. doi: 10.13703/j.0255-2930.20190316-k00034. Chinese. PMID 32100507
- [Background] Weijenborg PW, Cremonini F, Smout AJ, Bredenoord AJ. PPI therapy is equally effective in well-defined non-erosive reflux disease and in reflux esophagitis: a meta-analysis. Neurogastroenterol Motil. 2012 Aug;24(8):747-57, e350. doi: 10.1111/j.1365-2982.2012.01888.x. Epub 2012 Feb 6. PMID 22309489
- [Background] Yang J, Wang C. [Electroacupuncture at "Zusanli"(ST 36) can inhibit frequencies of transient lower esophageal sphincter relaxation induced by gastric distention in cats]. Zhen Ci Yan Jiu. 2011 Dec;36(6):423-7. Chinese. PMID 22379788
- [Background] Zachariah RA, Goo T, Lee RH. Mechanism and Pathophysiology of Gastroesophageal Reflux Disease. Gastrointest Endosc Clin N Am. 2020 Apr;30(2):209-226. doi: 10.1016/j.giec.2019.12.001. Epub 2020 Feb 5. PMID 32146942
- [Background] Zhang XP, Jia CS, Wang JL, Shi J, Zhang X, Li XF, Xu XK, Qin L, Zhang ML, Kang SG, Duan XD. [Acupoint catgut-embedding therapy: superiorities and principles of application]. Zhongguo Zhen Jiu. 2012 Oct;32(10):947-51. Chinese. PMID 23259283
- [Background] Zhu J, Guo Y, Liu S, Su X, Li Y, Yang Y, Hou L, Wang G, Zhang J, Chen JJ, Wang Q, Wei R, Wei W. Acupuncture for the treatment of gastro-oesophageal reflux disease: a systematic review and meta-analysis. Acupunct Med. 2017 Oct;35(5):316-323. doi: 10.1136/acupmed-2016-011205. Epub 2017 Jul 8. PMID 28689187
- [Background] Zou D, Chen WH, Iwakiri K, Rigda R, Tippett M, Holloway RH. Inhibition of transient lower esophageal sphincter relaxations by electrical acupoint stimulation. Am J Physiol Gastrointest Liver Physiol. 2005 Aug;289(2):G197-201. doi: 10.1152/ajpgi.00023.2005. Epub 2005 Apr 14. PMID 15831714
- [Result] Luo Z, Hu X, Chen C, Zhu L, Zhang W, Shen Y, He J. Effect of Catgut Embedment in Du Meridian Acupoint on Mental and Psychological Conditions of Patients with Gastroesophageal Reflux Disease. Evid Based Complement Alternat Med. 2020 Sep 22;2020:5415813. doi: 10.1155/2020/5415813. eCollection 2020. PMID 33029166
- [Derived] Trinh DT, Tran AH, Bui MP, Vuong NL. Thread-embedding acupuncture may improve symptom resolution in patients with gastroesophageal reflux disease: A randomized controlled trial. Integr Med Res. 2023 Sep;12(3):100971. doi: 10.1016/j.imr.2023.100971. Epub 2023 Jul 7. PMID 37637187